CLINICAL TRIAL: NCT06239597
Title: Effectiveness and Mechanisms of Lifestyle Intervention for College Students: Competence for Lifestyle Change, Occupational Balance, Perceived Health, and Well-being
Brief Title: Effectiveness and Mechanisms of Lifestyle Intervention for College Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: Ministry of Education, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ling-Hui Chang, Associate Professor, National Cheng Kung University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PMN1110332
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Lifestyle, Healthy
Keywords: lifestyle intervention; college student; online

STUDY DESIGN:
Intervention Model Description: an experimental group and a control group will be applied.
Who Masked: Participant
Masking Description: The intervention providers are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online lifestyle course (Experimental): 2 hours/session, one session/week, for 9 weeks. Online discussions, reflections, and activities are designed based on the Lifestyle Redesign literature and the health self-management knowledge.
  Interventions: Behavioral: occupation-based lifestyle intervention
- Control (Active Comparator): Ordinary college courses
  Interventions: Other: Other courses

INTERVENTIONS:
Behavioral: occupation-based lifestyle intervention — 9 week lifestyle course
  Arms: Online lifestyle course
Other: Other courses — Other courses in the same university, during the same academic years.
  Arms: Control

SUMMARY:
The goal of this trial is to test the effectiveness and learn about the mechanisms and effectiveness of lifestyle intervention for college students. The main questions it aims to answer are:

* Is the lifestyle course for college students effective in improving the skills and confidence for changing lifestyle, occupational balance, perceived health, as well as well-being for college students?
* What are the mechanisms between the course design and the students' learning?

Participants will join a 9-week online course that aims to facilitate college students to create health-promoting and satisfying habits and routines. Potentially a mixed format of online and in-person course design will be applied, depending on the university requirements and student feedback. Researchers will compare the experimental group and control group to see if the lifestyle tele-course improves college students' skills and confidence for changing lifestyle, occupational balance, perceived health, as well as well-being.

DETAILED DESCRIPTION:
1. Background:

   College students demonstrate a need for enhanced engagement in health-related lifestyles, including physical activities, nutritional behaviors, and stress management. In addition, past surveys reported that college students are frequently faced with adjustment problems in time management, a propensity for oversleeping, irregular sleep patterns, lack of life focus, ineffective study habits, academic stress, lack of motivation for studying, poor physical stamina, and easily experience fatigue in their functional arrangements. These lifestyle-related challenges can compromise health and quality of life. Although many college students have tried hard to "make changes" to their daily life, only some of them smoothly make the change.

   Our pilot study found that "Occupation and Health Promotion," a practice-oriented 8-week lifestyle course delivered by distance learning, could promote college students' skills and confidence for lifestyle change, occupational balance, and perceived-health. However, we also observed that the students did not consistently make behavioral changes in different lifestyle topics. Besides, some topics were perceived as more helpful, while others were not. Therefore, this study uses a systematic approach to explore the process of behavioral changes or no-changes, in order to look into the mechanism between the course design and the facilitated behavioral changes. In addition, the effectiveness shown in the pilot studies is expected to be replicated in this study.
2. Research purpose:

   1. To examine the effectiveness of the lifestyle course for college students, in terms of the skills and confidence for changing lifestyle, occupational balance, perceived health and well-being.
   2. To explore the mechanisms between the course design and the students' learning.
3. Research hypothesis:

   Intervention group will demonstrate greater efficacy in skills and confidence for changing lifestyle, occupational balance, perceived health and well-being compared to the control group.
4. Research Design:

   Mixed-method approach was selected. Three phases of the research protocol are as follows:
   1. Phase 1: Optimization of the course The optimization of the course will be grounded upon the detailed observations and documents of the course in the pilot studies, focus group of the participating students, one-on-one interview of college students, and expert reviews. Narrative analysis will be used to explore the process of behavioral changes, and the results will be triangulated with the Transtheoretical Model of Behavioral Changes, in order to improve the course design, such as effective teaching strategies and weekly teaching protocols.
   2. Phase 2: Effectiveness of the course The effectiveness of the course will be examined by non-randomized design with an experimental group and a control group. Questionnaires will be administered at pre-test, post-test, follow-up test after 2 months, follow-up test after 6 months. Sample size was calculated with G*Power 3.1.9.7. Attrition rate is estimated to be 87.5% at the second follow-up test. Consequently, 100 participants will be recruited in each group.

      The experimental group's intervention is an online course, potentially a mixed format of online and in-person, depending on the university requirements and student feedback; the control group participates in other university courses. The course of the experimental group consists of 100-minute weekly sessions for a total of nine weeks. The course is tailored to bolster students' ability to modify their lifestyles, thereby enriching their university experience with greater satisfaction and health. The course design is grounded in Experiential Learning, Lifestyle Redesign, self-management program, and the Transtheoretical Model of Behavioral Change, ensuring a comprehensive and practical learning experience.

      Self-rated online questionnaires will be used to assess motivation to behavioral changes, knowledge, attitude, skills, and self-efficacy for lifestyle change, occupational balance, health, as well as well-being. Descriptive analysis and two-way repeated-measures ANOVA will be conducted with IBM SPSS 17.0.
   3. Phase 3: Mechanisms of change Qualitative narrative analysis of the class materials, including group discussion records, self-reflection papers, and final reports, will be used to explore the mechanisms between the teaching strategies and the facilitated behavioral changes.
5. Expected contribution:

   1. This research will develop a distance lifestyle intervention approach which is effective in facilitating college students to gain competence in making lifestyle change, adopting a healthy lifestyle, as well as improving health and well-being.
   2. This research will contribute to the knowledge of concrete, feasible, and effective behavior change intervention targeting young adults, aiming at health promotion.
   3. Distance learning lifestyle courses can transcend spatial limitations, thereby enhancing student motivation to participate. Practical and executable lifestyle online courses will facilitate future health promotion for college students.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled college students

Exclusion Criteria:

* students who are unable to complete the questionnaires smoothly due to language barriers with Traditional Chinese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Stages of Change Ladder | Questionnaires will be administered at pre-test, post-test, follow-up test after 2 months, follow-up test after 6 months.
  The Stages of Change Ladder is a self-assessment 'readiness for action' scale, developed based on the Transtheoretical Model of Behavior Change. It assesses the respondent's self-rated readiness to change a specific problem or behavior, with participants choosing which step best represents their current thoughts or behavioral state. A higher score indicates greater readiness. For instance, 0 signifies no intention to change, while 10 indicates active behaviors are being taken.
Healthy Occupation and Lifestyle Competence Scale (HoLCS) | Questionnaires will be administered at pre-test, post-test, follow-up test after 2 months, follow-up test after 6 months.
  Measures the willingness for a healthy lifestyle (5 items) and the lifestyle adjustment skills (4 items). Using numerical rating scale scoring from 1 to 10, higher scores indicate higher levels of lifestyle competence. HoLCS demonstrated good content validity, good internal consistency, good convergent validity, and good construct validity based on confirmatory factor analysis.

SECONDARY OUTCOMES:
Occupational Balance Questionnaire 11-Chinese version (OBQ11_C) | Questionnaires will be administered at pre-test, post-test, follow-up test after 2 months, follow-up test after 6 months.
  Measures occupational balance, i.e., subjectively feeling that life consists of an appropriate amount and variety of occupations. It consists of 11 items, with a total score of 33. Each item is rated on a Likert scale for agreement with the statement: strongly disagree (0), disagree (1), agree (2), strongly agree (3). OBQ11-C has good expert validity (scale-level CVI = .93) and, with a sample of Taiwanese patients with depression, the questionnaire demonstrated good reliability, including internal consistency (Cronbach's α=0.898), test-retest reliability (ICC=0.818), and a four-point scale structure supported by Rasch analysis.
Self-perceived Health Scale | Questionnaires will be administered at pre-test, post-test, follow-up test after 2 months, follow-up test after 6 months.
  Refers to past research on self-perceived health, selecting three questions to inquire about overall self-perceived health, health compared to others, and satisfaction with overall health. It uses a 1 to 10 numerical rating scale, with higher scores indicating better perceived health. Based on students who took the course in the 2022, the three questions on self-perceived health demonstrated good internal consistency (Cronbach's α = .913)
Taiwanese Version of the World Health Organization-Five Well-Being Index (WHO-5-TW) | Questionnaires will be administered at pre-test, post-test, follow-up test after 2 months, follow-up test after 6 months.
  Measures subjective psychological well-being. It consists of five questions asking about the frequency of well-being status in the past two weeks, with higher scores indicating more frequent comfort: never (0), sometimes (1), less than half the time (2), more than half the time (3), most of the time (4), all the time (5). This scale has good clinical validity and is suitable for outcome evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Hui Chang, PhD, Study Chair — Department of Occupational Therapy, National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Participants were not requested to consent to the sharing of their data beyond the specific scope of this study. Consequently, in adherence to privacy and confidentiality considerations, we are unable to make their individual data available for external use.